CLINICAL TRIAL: NCT04851626
Title: Hypnotic Intervention for Women With Chronic Pelvic Pain: a Pilot Randomised Control Trial
Brief Title: Hypnotic Intervention for Women With Chronic Pelvic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Australia (Other)
Responsible Party: Principal Investigator, Tiffany Brooks, Principal Investigator, University of South Australia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202935
Record Dates: First submitted 2021-04-08; First posted 2021-04-20 (Actual); Last update posted 2021-04-20 (Actual); Status verified 2021-04

CONDITIONS: Chronic Pain; Pelvic Pain; Psychological; Hypnosis, Animal
MeSH Terms: conditions — Chronic Pain; Pelvic Pain; Immobility Response, Tonic

STUDY DESIGN:
Intervention Model Description: Pilot randomised controlled trial with 2 parallel study arms.
Masking Description: Masking not feasible for pilot design.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group - hypnotic intervention for persistent pelvic pain (Experimental): Participants underwent education about persistent pain and a 7 week 7 recording online hypnotic intervention. Women with persistent pelvic pain.
  Interventions: Other: Hypnotic intervention for persistent pelvic pain.
- Control group - waitlist control (Other): Control group of women with persistent pelvic pain no intervention completed assessment and concluding measures but did not undergo hypnotic intervention.
  Interventions: Other: Control group persistent pelvic pain no intervention.

INTERVENTIONS:
Other: Hypnotic intervention for persistent pelvic pain. — Education about persistent pelvic pain followed by 7 recordings of hypnosis intervention across 7 weeks accessed online through recordings.
  Arms: Intervention group - hypnotic intervention for persistent pelvic pain
Other: Control group persistent pelvic pain no intervention. — Control group no hypnotic intervention. Waitlist control.
  Arms: Control group - waitlist control

SUMMARY:
Objective: To establish whether the pilot online hypnosis design was well received by women with persistent pelvic pain and worthy of a full randomised control trial To establish whether hypnosis improves mental health outcomes, including anxiety, depression, life impact and catastrophizing, in women with chronic pelvic pain conditions.

DETAILED DESCRIPTION:
Design: Pilot Randomised Control Trial Methods: Twenty women with persistent pelvic pain completed assessment questionnaires and were recruited from a variety of social media sites related to persistent pelvic pain and randomly allocated to either control or hypnotic intervention groups. The intervention group completed a seven week online hypnotic intervention. The control group received no intervention. Both groups completed assessment and concluding questionnaires related to demographic information and the outcomes of interest. This included measures for anxiety, depression, pain, coping styles, pain related disability, pain catastrophizing and suggestibility. The results of the intervention and waitlist control groups were compared using linear mixed-effects modelling. Suggestibility was screened for at baseline using the Short Suggestibility Scale, and included in a secondary set of linear effects modelling.

ELIGIBILITY:
Inclusion Criteria:

* Meets criteria for persistent pelvic pain. Having experienced pain in the pelvic region below the umbilicus for over three months either beyond the healing time of a pathology or injury or without a diagnosed cause.
* Must be biologically female.
* Must be over the age of 18 years old.

Exclusion Criteria:

* Must not have a previously diagnosed or current mental health disorder involving dissociative states. Examples include diagnosed or current symptoms of Bipolar Type 1 or 2, psychotic disorders, untreated Post-Traumatic Stress Disorder.
* Must not reported current plan or intent to commit suicide.

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2020-11-02 (Actual); Primary Completion 2020-12-21 (Actual); Study Completion 2020-12-21 (Actual)

PRIMARY OUTCOMES:
Feasibility of hypnotic intervention according to qualitative responses from women with persistent pelvic pain. | 7 weeks
  Whether hypnosis was received well by women with persistent pelvic pain in the intervention group according to their qualitative responses during and after the study. Qualitative responses were collected in open text box format and analysed for themes using the thematic analysis software contained in the SurveyMonkey online software. There are no minimum, maximum or total scores as this was a free text response format.

SECONDARY OUTCOMES:
Impact on pain severity as indicated on a visual analogue scale (10 point). | 7 weeks
  Whether hypnotic intervention lead to significant differences in pain severity intervention group in comparison to controls. Pain severity was measured on a 10-point visual analogue scale. In terms of scores, 0 indicated no pain and 10 indicated the most severe pain possible. Higher scores indicated more pain severity. Minimum score is 0 and maximum potential score is 10.
Impact on depression scores on the Patient Health Questionnaire nine-item scale | 7 weeks
  Whether hypnotic intervention lead to significant differences in depression scores on the Patient Health Questionnaire nine-item scale in intervention group in comparison to controls.The scale has nine questions about depression symptoms, that are each scored on a scale of 0 (not at all) to 3 (nearly every day). The minimum score was 0 and the maximum score is 27, with higher scores meaning more depression symptoms present.
Impact on anxiety scores on the Generalised Anxiety Disorder scale seven-item | 7 weeks
  Whether hypnotic intervention lead to significant differences in anxiety score on the Generalised Anxiety Disorder 7-item scale for the intervention group in comparison to controls. The Generalised Anxiety Disorder seven-item has seven questions about anxiety symptoms scored from 0 (not at all) to 4 (every day). The minimum score in 0 and maximum score is 28, with higher scores indicating more anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Tiffany Brooks, Principal Investigator — University of South Australia
Locations (1):
- University of South Australia, Adelaide, South Australia, Australia

IPD SHARING:
Plan to Share IPD: No
Permission was only sought for participants in this study.

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-11-20): https://cdn.clinicaltrials.gov/large-docs/26/NCT04851626/Prot_SAP_000.pdf
  • Informed Consent Form (2020-11-20): https://cdn.clinicaltrials.gov/large-docs/26/NCT04851626/ICF_001.pdf